CLINICAL TRIAL: NCT07181577
Title: Sleep and Blankets
Acronym: SWAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Ali Amidi, Associate professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0367531; 1-10-72-90-25 (Other: The Regional Research Ethics Committees)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sleep Problems; Insomnia
Keywords: insomnia; sleep; RCT; blankets; actigraphy; sleep problems; sleep quality; young adults; sleep interventions; sleep disturbances; saliva; adolescents
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial (RCT) design with three parallel arms to evaluate the effects of a special blanket on sleep problems. Participants are randomly assigned to one of three groups.
  Group 1: receives Blanket A for home use over 4 weeks. Group 2: receives Blanket B for 4 weeks. Group 3 (observation group): receives no blanket during the same period but completes identical assessments.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Blanket A) (Experimental): Blanket A to be used in 4 weeks (Phase 1 - RCT) and the opportunity for additional 8 weeks (Phase 2 - open trial)
  Interventions: Device: Special blanket
- Group 2 (Blanket B) (Active Comparator): Blanket B to be used in 4 weeks (Phase 1 - RCT) and the opportunity for additional 8 weeks (Phase 2 - open trial)
  Interventions: Device: Different special blanket
- Group 3 (observational) (No Intervention): Sleep with their own blanket throughout the both Phase 1 and Phase 2

INTERVENTIONS:
Device: Special blanket — Special blanket to be used at home every night in 4 weeks (Phase 1 - RCT) and opportunity for additional 8 weeks (Phase 2 - open trial)
  Arms: Group 1 (Blanket A)
Device: Different special blanket — Different special blanket to be used at home every night in 4 weeks (Phase 1 - RCT) and opportunity for additional 8 weeks (Phase 2 - open trial)
  Arms: Group 2 (Blanket B)

SUMMARY:
Purpose

The primary aim of this research project is to evaluate whether a special blanket is an effective intervention for improving sleep among young people aged 16-24 with sleep disturbances. Sleep problems are increasingly common among Danish youth, with approximately one in five reporting significant sleep difficulties in the past 14 days. This trend has been rising steadily since 2010 and is mirrored internationally. Sleep disturbances are linked to a wide range of physical and mental health problems, including stress, anxiety, and depression, as well as negative effects on academic performance and social relationships. Early intervention is crucial to prevent chronic insomnia and poor mental health outcomes in adulthood.

Current treatments include specialized psychological therapies and medication. However, psychological therapies require extensive time and commitment, and medication carries risks of side effects, tolerance, and dependency, making non-pharmacological, safe, and accessible alternatives necessary. The special blanket is believed to promote relaxation through stimulation of the tactile and proprioceptive systems. Although promising in clinical and pedagogical contexts for certain populations (e.g., children with developmental disorders and adults with neurological conditions), there is limited scientific evidence regarding its efficacy and underlying mechanisms, particularly among youth with sleep disturbances.

Methods and Study Design

This project is a Phase 1 randomized controlled trial (RCT) assessing the effect of 4 weeks of using a special blanket on sleep problems among young people aged 16-24, as well as the impact on participants' mental and physical health. Additionally, the study investigates possible stress-related mechanisms involved in the use of the special blanket. Following the 4-week intervention, an open-label extension phase of 8 weeks (Phase 2) will explore continued use and acceptability of the blanket.

Eligible participants, screened for sleep problems, will be randomly assigned to one of three groups:

Group 1: receives a special blanket (Blanket A) for home use over 4 weeks.

Group 2: receives another special blanket (Blanket B) for 4 weeks.

Group 3 (observation group): no blanket provided but followed for 4 weeks to monitor changes in sleep problems.

The 4-week intervention phase (Phase 1) includes baseline (T1, week 0), mid-intervention (T2, week 2), and post-intervention (T3, week 4) online assessments. Sleep disturbances, physical and mental health, and stress-related mechanisms will be measured using validated questionnaires administered through REDCap. The first 40 participants in Groups 1 and 2 will additionally provide saliva samples and wear a circadian rhythm monitor (activity watch).

In Phase 2, participants in Groups 1 and 2 may continue using the blanket or revert to their usual bedding. At the end of Phase 2 (T4, week 12), follow-up questionnaires will assess sleep and user experience, including satisfaction, perceived benefits, barriers, and drawbacks of the blanket. Group 3 will then be offered a special blanket for an 8-week trial.

Participants The investigators aim to recruit 672 young people aged 16-24 with sleep problems.

Inclusion criteria are age 16-24 years and sleep problems measured by Insomnia Severity Index (score >10). Exclusion criteria are any underlying somatic, psychological, or neurological condition significantly affecting sleep quality; use of medications affecting sleep; pregnancy; shift work or night work; previous use of special blankets for sleep improvement and insufficient Danish language skills (questionnaires in Danish).

Significance and Relevance

The investigators anticipate that the findings will contribute to the current understanding of the non-pharmacological management of sleep problems, related mental and physical health outcomes, and underlying stress-related mechanisms of special blanket interventions. The results will be relevant to health professionals working with sleep problems, but also to adolescents and younger adults with sleep problems and their parents. New clinical guidelines on sleep problems in children and adolescents recommend non-pharmacological treatments as the first choice, specifically mentioning the potential efficacy of special blankets. The proposed project will help inform further development of such guidelines and related clinical practice. If special blankets are found to be effective in reducing insomnia, they could serve as an inexpensive, easily disseminated, and administered treatment with no known side effects, with the potential to greatly reduce the personal, as well as societal costs of insomnia.

DETAILED DESCRIPTION:
BACKGROUND Sleep problems are particularly common among adolescents and young adults, a developmental period characterized by biological, psychological, and social changes that increase vulnerability to insomnia. In Denmark, youth aged 16-24 report the highest prevalence of sleep difficulties, and similar trends are seen internationally. Short or disturbed sleep is linked not only to daytime fatigue, impaired academic performance, and social difficulties, but also to increased risk of stress-related disorders, anxiety, depression, and later chronic insomnia. Despite these risks, existing treatment options remain limited. Cognitive-behavioral therapy for insomnia (CBT-I) is effective but resource-intensive, while pharmacological treatments carry risks of side effects and dependency. Safe, accessible, and scalable non-pharmacological alternatives are urgently needed.

Special blankets represent one such potential intervention. These blankets can be designed to stimulate tactile and proprioceptive systems, which may reduce hyperarousal, promote relaxation, and regulate stress-related mechanisms. Preliminary observations suggest beneficial effects on sleep initiation and maintenance, as well as reductions in anxiety and stress. However, robust randomized controlled trials (RCT) in general youth populations with clinically relevant insomnia are lacking.

AIMS AND HYPOTHESES

Primary aim Aim 1: To test the efficacy of different blankets on insomnia severity (primary outcome) in adolescents and young adults with insomnia.

Exploratory aims Aim 2: To test the effect of different blankets on actigraphy-based sleep (sleep efficiency, total sleep time and wake after sleep onset) in a sub-group of adolescents and young adults.

Aim 3: To explore the effect of different blankets on self-report measures of mental and physical health and well-being (i.e., stress, depression, anxiety, cognition, daytime sleepiness, health status and quality of life) in adolescents and young adults.

Aim 4: To explore the effect of different blankets on potential stress-related mechanisms (i.e., the diurnal cortisol response and self-reported pre-sleep arousal) and to test for potential mediation of the effect of special blankets on insomnia severity.

Aim 5: To explore the continued use of different blanket for 8 weeks after intervention completion and to track associated changes in insomnia severity and self-reported mental health and physical well-being in an open trial design.

METHODS

The present project aims to fill this knowledge gap through a rigorous, two-phase study design. In Phase 1, a randomized controlled trial (RCT) will test the efficacy of different special blankets compared with an observation group receiving no blanket. Eligible participants will be young people aged 16-24 with clinically relevant sleep problems, defined as an Insomnia Severity Index (ISI) score >10. After baseline screening and consent, participants will be randomized via REDCap into one of three groups:

Group 1: receives Blanket A for home use over 4 weeks.

Group 2: receives Blanket B for 4 weeks.

Group 3 (observation group): receives no blanket during the same period but completes identical assessments.

Assessments will take place at baseline (week 0), mid-intervention (week 2), and post-intervention (week 4). Primary outcomes will be insomnia severity and sleep quality, assessed by validated questionnaires. Secondary outcomes include mental health indicators (stress, anxiety, depressive symptoms), physical health, and well-being. To explore potential mechanisms, the first 40 participants in Groups 1 and 2 will also provide salivary cortisol samples and wear actigraphy devices to measure circadian rhythm and sleep-wake patterns.

In Phase 2, an open-label extension phase, participants in Groups 1 and 2 may continue using their blanket or revert to regular bedding for an additional 8 weeks. At week 12, follow-up questionnaires will assess long-term sleep outcomes, user experience, satisfaction, and perceived barriers. Participants from the observation group will then be offered the opportunity to try a special blanket for 8 weeks, ensuring equal access.

The investigators plan to recruit 672 participants, which will provide sufficient statistical power to detect clinically meaningful effects while accounting for potential dropout. Inclusion criteria are age 16-24 years and ISI >10. Exclusion criteria include significant somatic, psychiatric, or neurological disorders affecting sleep; ongoing use of medications influencing sleep; pregnancy; shift or night work; prior use of special blankets for sleep; and insufficient Danish language proficiency to complete questionnaires.

SIGNIFICANCE AND RELEVANCE This project will be the first large-scale, randomized evaluation of special blankets in a general youth population with insomnia symptoms. By integrating subjective measures, objective circadian monitoring, and biological stress markers, the study will not only test efficacy but also shed light on underlying mechanisms. Results will have direct clinical relevance: recent guidelines for managing sleep problems in children and adolescents emphasize non-pharmacological approaches and highlight the potential of special blankets as a first-line option. If proven effective, special blankets could represent a safe, inexpensive, and easily disseminable intervention with the potential to substantially reduce the personal and societal burden of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 16 and 24 years old
* Participants must have a score on the Insomnia Severity Index (ISI) above 10.

Exclusion Criteria:

* Presence of neurological disorders known to influence or be related to poor sleep including affective disorders and diagnosed medical sleep disorders (e.g., sleep apnea, narcolepsy)
* Circulatory or respiratory disease
* Pregnancy, shift or night work
* Prior use of special blanket (within the past five years)
* Insufficient Danish proficiency.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 672 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  Insomnia Severity Index (ISI) will be used to assess the severity of insomnia symptoms. The ISI is a brief self-report instrument consisting of seven items that evaluates the severity of sleep-onset, sleep maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and level of distress caused by the sleep problem. This corresponds in part to the diagnostic criteria of insomnia. Zero is the minimum value and equivalent to no insomnia and 28 is the maximum value and indicates clinical insomnia in severe degree.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Pittsburg Sleep Quality Index (PSQI) will be used in order to measure subjective sleep quality. It consists of 19 self-rated items and has high internal consistency (Cronbach's α = 0.83) and test-retest reliability (r = 0.85). The minimum score is 0 and the maximum score is 21, with higher scores indicating poorer sleep quality.
Actigraphy-based sleep | Baseline (T1) and Week 4 (T3)
  ActTrust 1 (Condor Instruments, São Paulo, Brazil) will be used to measure rest/wake activity for 8 days at two timepoints in a subgroup (n=80). In addition to sleep/wake activity, ActTrust records information about amount and duration of ambient light and wrist temperature, allowing analyses of whether observed effects are related to group-differences in temperature. Extracted sleep variables include sleep onset latency (SOL), total sleep time (TST), sleep efficiency (SE), and wake after sleep onset (WASO). To help edit actigraphy data, participants will complete a sleep diary during this period, giving information about bedtime, time spent falling asleep, wake up time, rise time, estimated number of awakenings and self-rated sleep quality.
Diurnal salivary cortisol | Baseline (T1) and Week 4 (T3)
  Diurnal salivary cortisol will be measured in a subgroup of participants (n = 80, 40 from each of groups 1 and 2) at two different time points. At each of these time points, participants will be instructed in home-based self-collection of 5 daily saliva samples for two consecutive days. The daily samples will be collected at personal waking (#1); 30 min. after waking (#2); 45 min. after waking (#3); between 4 and 6pm (#4); and at bedtime (#5). This sampling schedule allows for the assessment of both diurnal cortisol patterns and Cortisol Awakening Response (CAR) estimation. Samples will be collected in labelled Sarstedt salivettes and stored in sealable dark plastic bags to protect from sun exposure. Collection time will be written on the salivette by participants.
Stress | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Depression | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Patient Health Questionnaire-9 (PHQ-9) is a brief, self-administered tool used to screen for and assess the severity of depression in patients. It consists of nine questions about depressive symptoms experienced over the past two weeks, with answers scored on a 0-3 scale to determine the severity of depression. A total score is calculated, with higher scores indicating greater severity. The minimum score is 0 and the maximum score is 27.
Anxiety | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Generalised Anxiety Disorder Assessment (GAD-7) is a brief measure for symptoms of anxiety, based on the generalised anxiety disorder (GAD) diagnostic criteria described in the Diagnostic and Statistical Manual of Mental Disorders (DSM). A raw score (from 0 to 21) is presented as well as a percentile rank based on a normative community sample of age-related peers. Higher scores indicate higher levels of anxiety.
Cognitive impairment | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Cognitive Failures Questionnaire (CFQ) measures how often people experience cognitive failures. Examples of cognitive failures include: forgetfulness, distractibility, and poor cognitive or behavioral performance that may be related to stress, mental health issues, physical health issues, or neurocognitive disorders (NOT due to ability). Respondents answer how often they experience the cognitive symptoms listed (e.g., "Do you find you forget your appointments?") on a scale from "Never" to "Very often". The CFQ contains 25 questions scored on a 5-point Likert scale from 0 ("Never") to 4 ("Very often"). A total score is obtained by summing the item responses and ranges from 0 to 100. Higher scores suggest higher frequency of cognitive failures.
Daytime sleepiness | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.
  0-5 Lower Normal Daytime Sleepiness 6-10 Higher Normal Daytime Sleepiness 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness 16-24 Severe Excessive Daytime Sleepiness
Health related quality of life | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Scores range from 0-100, with higher scores indicating better health (less pain, more function).
Mental well-being | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The WHO-5 is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.
  The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Background information | Baseline (T1)
  Information on sociodemographic factors and comorbidity will be self-reported by all participants
Health-related behaviors | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  Information about drugs, smoking, exercise, medical use, use of digital devices, nutrition etc.
Sleep arousal | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  The Pre-Sleep Arousal Scale (PSAS) is a validated and reliable self-report measure that will be used to assess evening pre-sleep arousal. It has been widely used in research as a reliable marker for cognitive and somatic arousal including in younger adults. On the Pre-Sleep Arousal Scale (PSAS), scores range from 16 to 80, with higher scores indicating greater pre-sleep arousal.
Circadian predispositions | Baseline (T1), week 2 (T2), Week 4 (T3), week 12 (T4). To measure change across timepoints.
  Circadian predispositions will be assessed using the 5-item self-rated reduced version of the Morningness-Eveningness Questionnaire (MEQr), which measures whether a person's peak alertness is in the morning or evening. The Morningness-Eveningness Questionnaire, Revised Short Form (rMEQ) is a shortened, five-item version of the original Horne and Östberg MEQ, developed to quickly assess an individual's chronotype (whether they are a morning or evening type) with good reliability and validity. The scores are summed, with a higher total score typically indicating morningness and a lower score indicating eveningness.
  Scores typically range from 4 or 5 to 25 or 27, depending on the specific scoring methodology used. The sum total classifies individuals into categories:
  Evening types (e.g., scores 4-10), Intermediate/Neither types (e.g., scores 11-18), Morning types (e.g., scores 19-25).
Credibility/Expectancy | Baseline (T1)
  The Credibility/Expectancy Questionnaire will be used to assess treatment credibility and outcome expectancy. The measure was developed for clinical studies to measure treatment expectancy and rationale credibility. A minimum score of 6 and a maximum score of 54 for the total score, when all items are summed. Higher scores on both subscales and the total score reflect greater perceived treatment credibility and higher outcome expectancy.
Questionnaire on evening activity, adherence and user experience | Week 2 (T2), Week 4 (T3), Week 12 (T4)
  Participants will also be asked to respond to questions about adherence and user experience of the assigned blanket in order to assess adherence, treatment satisfaction and potential barriers to use of weighted blankets. An extended version with open-ended questions about their experience with the blankets will be used during the follow-up assessment at the end of the open-trial period (T4).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology and Behavioural Sciences, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Will not be shared